CLINICAL TRIAL: NCT07095153
Title: Examining the Effects of a Neuroathletic Training Program on the Physical, Cognitive, and Performance Abilities of Judokas
Brief Title: Effects of Neuroathletic Training on Judokas' Physical, Cognitive, and Performance Abilities
Acronym: NAT-Judo
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Collaborators: Saglik Bilimleri Universitesi (Other); Igdir University (Other)
Responsible Party: Principal Investigator, BİNNAZ BOZKURT AKPULAT, Lecturer and PhD Candidate, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IGDU-EC-19-3-2025
Record Dates: First submitted 2025-07-14; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Neuroathletic Training; Exercise; Athletic Performance
Keywords: Neuroathletic training; Judo; Physical fitness; Cognitive performance; Sport performance; Exercise therapy
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Two-arm randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The outcome assessors and data analysts will be blinded to group allocation. Participants and intervention providers will not be blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuroathletic Training Group (Experimental): Within the scope of this study, the intervention group will undergo a Neuroathletic Training (NAT) protocol, performed three times per week over eight weeks. The program begins with 1 set of 30 seconds with 10 seconds of rest during the first two weeks, with the number of sets increasing every two weeks. Each training session includes 6 to 8 different exercises. The selected exercises target cognitive-neuromotor skills such as visual tracking, target following, shifting focus, decision-making, fall reflex, balance adaptation, motor coordination, and spatial perception. This program is integrated into the classical judo training and is limited to a total duration of 20 to 25 minutes per session.
  Interventions: Behavioral: Neuroathletic Training (NAT)
- Control Group (Other): Participants in the control group will perform only the classical judo training protocol throughout the study. This training is based on the training plans and technical development programs developed by the Turkish Judo Federation for the 10-18 age group.
  Interventions: Behavioral: Routine Judo Training

INTERVENTIONS:
Behavioral: Neuroathletic Training (NAT) — The intervention group will undergo an 8-week Neuroathletic Training program, conducted three times a week. The program consists of exercises designed to enhance visual-motor coordination, reaction time, balance, and proprioception, integrated with classical judo training. Each session lasts approximately 20-25 minutes and includes 6 to 8 different exercises targeting cognitive and neuromotor skills.
  Arms: Neuroathletic Training Group
Behavioral: Routine Judo Training — The control group will continue with their usual judo training program, which follows the training plans and technical development programs set by the Turkish Judo Federation for athletes aged 10-18. This program focuses on maintaining and improving existing technical, tactical skills, physical conditioning, and sports culture without any additional neuroathletic training interventions.
  Arms: Control Group

SUMMARY:
The primary objective of this project is to comprehensively investigate the effects of the Neuroathletic Training (NAT) approach, integrated into the routine training program, on the physical fitness, cognitive skills, and sports performance of judokas aged 10 to 18 years. This study is designed as a randomized controlled trial involving 40 judokas randomly assigned to either the NAT group or the control group. The NAT program, implemented over eight weeks, includes exercises targeting visual-motor coordination, reaction time, balance, and proprioception. Outcome measures such as reaction time, agility, balance, flexibility, proprioception, attention, grip strength, and judo-specific physical fitness will be assessed using a pre-test and post-test design. The results are expected to contribute to the development of a novel training model aimed at enhancing judo performance and to provide original insights into the effects of neuroathletic training in sports sciences. Additionally, the NAT protocol aims to improve not only physical fitness parameters but also cognitive domains such as mental flexibility, decision-making speed, and concentration by enhancing neuromotor control parameters including balance, coordination, reaction time, and attention.

DETAILED DESCRIPTION:
This study is a randomized controlled experimental design to be conducted on athletes aged 10 to 18 who regularly train in judo at the Iğdır Provincial Directorate of Youth Services and Sports. A total of 40 judokas will be homogeneously assigned to intervention and control groups using stratified randomization, and demographic data such as age, gender, height, weight, judo experience, and dominant side will be recorded.

The intervention group will undergo a neuroathletic training (NAT) protocol three times a week for eight weeks, while the control group will continue only with routine judo training. The NAT program consists of exercises aimed at improving visual-motor coordination, reaction time, balance, and proprioception, integrated with judo techniques to enhance motor outputs. The duration and number of sets of exercises will gradually increase over the weeks, with each session covering 6 to 8 different cognitive and neuromotor skills.

Pre-test and post-test measurements will be conducted using a comprehensive set of tools, including Judogi Isometric and Dynamic Barfiks Tests to assess judo-specific endurance and upper extremity strength, the Central Nervous System Vital Signs (CNSVS) computerized neuropsychological test battery to evaluate cognitive functions, the Sit and Reach Test for flexibility, hand dynamometer for grip strength, Single-Leg Stance Test for static balance, Y Balance Test for dynamic balance, Illinois Agility Test for rapid direction change and agility, Light Trainer system to measure reaction time, hand-eye and foot-eye coordination and reactive agility, and shoulder joint position sense assessment for proprioception. All assessments will be performed in a double-blind manner by two physiotherapists with five years of experience. The collected data will be anonymized and analyzed by an independent statistician who is blinded to group allocation.

Statistical analyses will be performed using SPSS 25.0 software; data distribution will be evaluated with the Shapiro-Wilk test. Paired and independent samples t-tests will be applied for normally distributed variables, while Wilcoxon and Mann-Whitney U tests will be used for non-normally distributed data. The significance level will be set at p < 0.05, and effect sizes will be calculated to assess the strength of the findings.

This study aims to comprehensively investigate whether neuroathletic training is effective in improving both the physical and cognitive performance of young judokas. The findings are expected to contribute to the development of training programs tailored to the developmental needs of children and youth athletes, as well as to enhance performance and reduce injury risk in complex sports such as judo.

Furthermore, this study is conducted under the supervision of Prof. Dr. Necmiye Ün Yıldırım, the thesis supervisor, and assisted by Assoc. Prof. Dr. Çağlar Soylu, both affiliated with the University of Health Sciences. The principal investigator is Binnaz Bozkurt Akpulat, a PhD candidate at the University of Health Sciences and a lecturer at Iğdır University.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 10 and 18 years
* Practicing judo regularly for at least 1 year
* Attended a minimum of 3 training sessions per week for the last 6 months
* Holding an active competitive license
* Medically cleared for sports participation
* No musculoskeletal restrictions that limit physical activity
* No diagnosed neurological or vestibular disorders
* Cognitive ability to understand and follow test procedures
* Written informed consent provided by parent/legal guardian (for participants under 18)
* Commitment to regular participation throughout the study duration

Exclusion Criteria:

* Individuals diagnosed with attention deficit, hyperactivity disorder, or difficulty maintaining attention during training
* Individuals using medications targeting balance, visual, or vestibular systems
* Participation in any other scientific study simultaneously
* Currently receiving psychiatric treatment or regular use of psychiatric medication
* Previous participation in neuroathletic or similar neuromotor training programs
* Individuals who actively resist or deliberately sabotage the NAA protocol
* Missing two or more measurement or training sessions during the study
* Refusal to comply with the protocol or failure to complete surveys/tests
* Participants whose parents/guardians express concerns or refuse approval during the consent process
* Behaviors that may jeopardize study sustainability or data integrity

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Reaction Time | 1 month
  Reaction time is an important performance indicator that reflects the speed of information processing and the ability to respond to stimuli in cognitive and perceptual processes. In this study, the Light Trainer application will be used to assess reaction time.
  Light Trainer operates with a wireless system consisting of eight LED lights. These lights are equipped with sensors that are activated by proximity or touch. The application is used to measure performance components such as agility, speed, coordination, and reaction time.
  Reaction time is measured in milliseconds (ms). In healthy individuals, this time typically ranges between 250-400 ms, while trained athletes are generally expected to perform below 250 ms, due to enhanced sensory processing and faster neuromuscular responses.
Reactive Agility | 1 month
  Reactive agility will be assessed using the Light Trainer system. The test begins when the athlete touches the centrally located LED light with their hand. Six LED lights, placed on cones at a height of 40 cm, light up in a random sequence. The athlete must identify the lit LED, quickly run to the corresponding cone, pass through a designated 20 cm area around the light using their preferred hand, and return to the base light. Reactive agility performance is recorded as the time interval between the activation of the first LED and the deactivation of the last LED.
  According to normative data, this time typically ranges between 5 and 10 seconds in healthy young adults. In experienced athletes, the performance time is generally around 4 to 6 seconds. Times are recorded in seconds according to the nature of the test.
Single Leg Stance Test | 3 weeks
  This test is applied to evaluate static balance. The athlete is instructed to stand on one foot with eyes closed and the knee flexed approximately at 90 degrees. The athlete is expected to maintain balance throughout the test duration. The time is measured with a stopwatch during each trial, and the test is repeated three times in total. The average of the three recorded times reflects the athlete's static balance performance.
Y Balance Test | 3 weeks
  This test will be used to evaluate dynamic balance of the lower and upper extremities. The setup consists of three measuring tapes arranged in a "Y" shape with 120° angles between them.
  For the lower extremity, the athlete will stand on one foot at the center of the tapes and reach as far as possible with the other foot in the anterior, posteromedial, and posterolateral directions. Leg length will be measured from the anterior superior iliac spine (ASIS) to the medial malleolus. The composite score will be calculated by summing the three reach distances, dividing by three times the leg length, and multiplying by 100.
  For the upper extremity, the athlete will stand on one hand at the center of the tapes and reach as far as possible with the other hand in the medial, inferolateral, and superolateral directions. Arm length will be measured from the seventh cervical vertebra (C7) to the tip of the middle finger. The composite score will be calculated similarly.
Central Nervous System Vital Signs (CNSVS) - Cognitive Function Assessment | 6 weeks
  The Central Nervous System Vital Signs (CNSVS) computerized neuropsychological test battery will be used to assess individuals' cognitive functions. The test is completed on a computer via a link sent by email and takes approximately 30-40 minutes. Detailed results are provided upon completion.
  CNSVS consists of seven subtests measuring cognitive domains such as executive functions, memory, attention, reaction time, and processing speed. These yield 11 domain scores and one neurocognitive index (NCI) score.
  NCI scores are interpreted as follows: above 110 indicates high cognitive capacity, 90-110 normal, 80-89 below normal, and 70-79 low cognitive capacity.

SECONDARY OUTCOMES:
Judogi Isometric Pull-Up Test (Upper Body Strength and Endurance) | 2 weeks
  Athlete holds two judogi ropes suspended from a bar and maintains an isometric pull-up (elbows maximally flexed) for as long as possible. Maximum hold time is recorded in seconds. Various normative values exist for the Judogi Isometric Pull-Up Test. Elite male judokas typically maintain the isometric hold for about 35 seconds, while non-elite judokas usually perform between 15 and 25 seconds.
Judogi Dynamic Pull-Up Test | 2 weeks
  The athlete holds judogi ropes suspended from a bar with hands facing forward and elbows fully extended. The athlete moves the elbow joint from full extension to full flexion repeatedly until fatigue. The highest number of repetitions achieved is recorded. Various normative values exist for the Judogi Dynamic Pull-Up Test. Elite male judokas typically perform around 12 repetitions, while non-elite judokas usually perform between 3 and 7 repetitions.
Sit and Reach Test | 2 weeks
  This test will be used to assess trunk and lower limb flexibility in children. The individual will sit with legs extended, placing the soles of the feet on the sit-and-reach box, and reach forward along a ruler while keeping the knees extended. The edge of the box will be considered zero; forward reaches will be recorded as positive values and backward movements as negative values. The test will be repeated three times, and the highest value in centimeters will be recorded.
Hand Grip Strength | 2 weeks
  Hand grip strength will be measured in kilograms (kg) using a hand dynamometer. The athlete will stand and grasp the dynamometer with the elbow fully extended. The arm and hand will not touch the body, and the athlete will apply maximal isometric grip force without moving the arm. This test, known for its high reliability, will be used in clinical research.
Illinois Agility Test | 2 weeks
  The Illinois Agility Test will be used to assess athletes' ability to change direction quickly and their agility. The test course will be set up on a judo mat, measuring 5 meters wide and 10 meters long, with four cones placed in a straight line at 3.3-meter intervals in the middle section.
  Athletes will start the test lying face down at the starting line, with their hands placed shoulder-width apart touching the ground. The test time will be recorded in seconds using a stopwatch. The test involves approximately 40 meters of straight running and 20 meters of slalom running, including 180° turns every 10 meters.
  Before the test, athletes will be familiarized with the course and allowed to perform 2-3 low-speed practice runs. This test is validated for reliability and applicability in adolescent and adult populations.
Hand-Eye and Foot-Eye Coordination | 1 month
  The Light Trainer system will be used to assess upper extremity hand-eye coordination and reaction speed. The athlete will stand in front of a table 80 cm high. Four spotlights will be arranged on the table in a row, spaced 30 cm apart. The athlete will try to touch as many lit spots as possible with their palm or fingers within 30 seconds. Two trials will be conducted for each hand, and the highest number of touches will be recorded.
  The Light Trainer system will also be used to evaluate lower extremity foot-eye coordination and reaction speed. The athlete will stand in front of four spotlights arranged in a row, spaced 30 cm apart. The athlete will try to touch as many lit spots as possible using the ball of their foot within 30 seconds. Two trials will be conducted for each foot, and the highest number of touches will be recorded.
  In both tests, the goal is to deactivate the lights as quickly and accurately as possible.
Proprioception Assessment | 3 weeks
  Joint position sense (JPS) test will be used to measure proprioceptive sense in the shoulder. The athlete will lie supine and position the arm at 90° abduction with 45° and 80° external rotation angles. The examiner will passively place the arm at the target angle and hold it for 5 seconds, then return it to the starting position. The athlete will actively reproduce the target angle and say "Done" when they believe the position is matched. Three trials will be performed for each angle and extremity. Absolute error score will be calculated as the average difference between the target and reproduced angles. The error score is measured in degrees (°).

CONTACTS AND LOCATIONS:
Overall Officials: Binnaz BOZKURT AKPULAT, PhD Cand., Principal Investigator — Igdir University; Necmiye ÜN YILDIRIM, Professor, Study Chair — Saglik Bilimleri Universitesi; Çağlar SOYLU, PhD, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Iğdır Provincial Directorate of Youth Services and Sports, Iğdır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data may be shared upon reasonable request and with appropriate data use agreements, following ethical approvals.